CLINICAL TRIAL: NCT05092321
Title: Exploration of Aquatic Therapy in Children With Autism and Their Families
Brief Title: Aquatic Therapy for ASD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: Franklin County Board of Developmental Disabilities (Unknown)
Responsible Party: Principal Investigator, Erika Kemp, Assistant Professor, Clinical, Ohio State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019J0204
Record Dates: First submitted 2021-09-16; First posted 2021-10-25 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Aquatic Occupational Therapy (Experimental): Group-based aquatic occupational therapy with 1:1 swim buddy for safety.
  Interventions: Behavioral: Aquatic Occupational Therapy

INTERVENTIONS:
Behavioral: Aquatic Occupational Therapy — Group of 4-8 children, paired with a swim buddy. Intervention techniques including discrete teaching, motor shaping, behavioral management, therapeutic relationship and individualized goals.

SUMMARY:
This is an aquatic occupational therapy group for children between the ages of 3-12 that have an autism diagnosis. Intervention will focus on increasing the child's safety swim skills.

DETAILED DESCRIPTION:
Information will be collected from participants' guardians during an intake visit regarding a child's sensory processing deficits, movement abilities and exposure to swim skill instruction prior to the group. The group will provide swim instruction using the Halliwick approach to learning swim skills as well as other occupational therapy techniques such as shaping, therapeutic relationship and behavior management. Groups will have a minimum ratio of 1 staff to every 2 children, with the possibility of 1:1 ratio most days. There will be a certified lifeguard present at all times. Qualitative interviews and a follow up survey will be conducted with parents (ages 18+) to determine impact on families and individual participants. Swim skills will be tracked at each session via goal attainment scaling and daily documentation. Descriptive and correlational statistics will be completed as well as coding of interview and survey data. Participants can participate for one, 10 week session, or will have the option to participate in additional 10 week sessions until child participants top out on the WOTA or plateau in progress of swim skills.

ELIGIBILITY:
Inclusion Criteria:

* pre-existing diagnosis of autism spectrum disorder from a medical professional
* family interest in swimming

Exclusion Criteria:

* ventilation system for breathing such as trachea not capped

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2021-09-14 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
Change in swim skills | baseline, pre-intervention; immediately after the intervention
  Change in swim skills measured with Water Orientation Test-Alyn; higher scores mean a better outcome. Minimum score is 0, maximum is 27
Change in individualized goals | immediately after the intervention
  Goal Attainment Scaling to track change in other swim performance skills not measured above. Scores for each goal range from -2 (regression) to +2 (2 levels more than anticipated). A higher score indicates improvement.
Change in parent comfort | baseline pre-intervention; immediately after the intervention
  Custom questionnaire using 5 point Likert scale regarding comfort and importance of water participation for the child. A higher score indicates increased parent comfort, which is the desirable direction.
Parent perspective | one time after 8 hours of intervention have been provided to the child participant
  qualitative interview regarding parent perspective of the the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Erika Kemp, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
De-identified data may be shared with other researchers.